CLINICAL TRIAL: NCT04076423
Title: A Phase IV, Multicenter, Open and Randomized Study to Assess the Impact of the Change From Antiretroviral Treatment From Dual Therapy to Triple Therapy on Inflammation in Patients With Type 1 HIV Infection. InSTINCT Study
Brief Title: A Phase IV Study to Assess the Impact of the Change of Antiretroviral Treatment From Dual Therapy to Triple Therapy on Inflammation in Patients With HIV Infection
Acronym: InSTINCT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundacion SEIMC-GESIDA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GeSIDA 10918
Record Dates: First submitted 2019-08-27; First posted 2019-09-03 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-06

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Dual Anti-Platelet Therapy

STUDY DESIGN:
Intervention Model Description: Comparator: the patient will continue taking the dual therapy. Experimental: the patient Will beging to take triple therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm: (Experimental): they will take 1 tablet (50 mg BIC + 200 mg FTC + 25 mg TAF), orally, once a day, from the moment of randomization.
  Interventions: Drug: Triple therapy
- Comparator arm (Active Comparator): they will take 1 tablet of 50 mg of DTG orally, once a day + 1 tablet of 300 mg of 3TC orally, once a day, from the randomization moment.
  Interventions: Drug: Dual Therapy

INTERVENTIONS:
Drug: Dual Therapy — DTG + 3TC
  Arms: Comparator arm
Drug: Triple therapy — BIC / FTC / TAF
  Arms: Experimental arm:

SUMMARY:
242 patients (121 patients in each of the two treatment arms) will be included with a confirmed diagnosis of HIV-1 infection and with a stable antiretroviral treatment during more than 48 weeks with dual therapy (DTG + 3TC)

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 18 years
* Confirmed and documented diagnosis of HIV-1 infection
* Virological suppression of more than 48 weeks (confirmed with HIV RNA <50 copies / ml). The determination of the CV of a routine prior analysis of ≤ 12 weeks prior to signature of consent.
* ART in stable dual therapy (> 48 weeks) with DTG + 3TC
* Signed informed consent
* Negative pregnancy test in urine or blood

Exclusion Criteria:

* Inability to obtain written informed consent to participate in the study
* Pregnant or breastfeeding women or those who intend to become pregnant during the study period and do not undertake to use proven contraceptive methods.
* Any suspicion or confirmation of resistance to TAF, 3TC, FTC, DTG or BIC. In case of have a study of baseline resistance mutations prior to the start of ART has to rule out resistance to investigational drugs.
* Patients with hypersensitivity to any excipient used with TAF, FTC, DTG or BIC
* Any chronic autoimmune or inflammatory disease
* Use of immunomodulatory or immunosuppressive agents, including steroids Chronic treatment with aspirin, statins and other anti-inflammatory agents
* Any acute infection in the last 2 months
* Estimated glomerular filtration rate (TFGe) <30 mg / ml / m2 measured by any of the formulas available. The determination of the TFGe of a previous routine analysis of ≤ 12 weeks prior to signing the consent is allowed
* Contraindication for the use of TAF
* Clinical condition of the patient in rapid deterioration or the investigator considers that there is no reasonable hope that the patient will finish the study
* Simultaneous participation in another clinical trial or research study that requires the need of treatment with other drugs outside the study or interfere with the visits of the same.
* Any situation that, in the opinion of the investigator, may interfere with the patient's ability to meet the treatment schedule and protocol evaluations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2024-01-16 (Actual)

PRIMARY OUTCOMES:
sCD14 | Screening, basal, week 23, week 24, week 47, week 48, week 95 y week 96
  Changes in sCD14 concentration

SECONDARY OUTCOMES:
Changes in PCR-us | Screening, basal, week 23, week 24, week 47, week 48, week 95 y week 96
  Inflammation (IL-6 signaling pathways):
Changes in sCD163 | Screening, basal, week 23, week 24, week 47, week 48, week 95 y week 96
  Monocyte / macrophage activation
Changes in quinurenine / tryptophan ratio | Screening, basal, week 23, week 24, week 47, week 48, week 95 y week 96
  IDO-1 induction
Changes in Dimer D | Screening, basal, week 23, week 24, week 47, week 48, week 95 y week 96
  Coagulation
Changes in CD4/CD8 ratio | Screening, basal, week 23, week 24, week 47, week 48, week 95 y week 96
  Inmunoactivation
Changes in CD4+ | Throughout all the study, an average of 100 weeks
Changes in viral suppression rates | Throughout all the study, an average of 100 weeks
Longitudinal trajectories of plasma biomarkers | Throughout all the study, an average of 100 weeks
  The differences in the trajectories of soluble inflammatory markers by comparing the slopes of each biomarker between treatment arms. Longitudinal changes in each biomarker will be compared using linear or non-linear mixed models with random intercepts, depending on the normality of the data.
Longitudinal trajectories of CD4/CD8 ratio | Throughout all the study, an average of 100 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Santiago Moreno, MD, Principal Investigator — Hospital Univ. Ramón y Cajal; Sergio Serrano, MD, Principal Investigator — Hospital Univ. Ramón y Cajal
Locations (18):
- Spain (18):
  - Hospital San Pedro, Logroño, La Rioja
  - Hospital Universitario Príncipe de Asturias, Alcalá de Henares, Madrid
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Hospital de Bellvitge, Barcelona
  - Hospital Univ. Vall D'Hebron, Barcelona
  - H. General Universitario Guadalajara, Guadalajara
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Fundación Jimenez Diaz, Madrid
  - Hospital Univ. La Paz, Madrid
  - Hospital Univ. Ramón y Cajal, Madrid
  - Hospital Virgen de las Nieves, Malá
  - Hospital Virgen de la Victoria, Málaga
  - H. General Universitario Reina Sofía, Murcia
  - Hospital Univ. Virgen del Rocio, Seville
  - H. Universitario y Politécnico La Fe, Valencia
  - Hospital Univ. Clínico de Valencia, Valencia
  - Hospital Univ. Lozano Blesa, Zaragoza

REFERENCES:
- [Derived] Saborido-Alconchel A, Serna-Gallego A, Trujillo-Rodriguez M, Munoz-Muela E, Alvarez-Rios AI, Lozano C, Llaves-Flores S, Espinosa N, Roca-Oporto C, Herrero M, Sotomayor C, Gutierrez-Valencia A, Lopez-Cortes LF. Long-term effects on immunological, inflammatory markers, and HIV-1 reservoir after switching to a two-drug versus maintaining a three-drug regimen based on integrase inhibitors. Front Immunol. 2024 Jul 11;15:1423734. doi: 10.3389/fimmu.2024.1423734. eCollection 2024. PMID 39055703